CLINICAL TRIAL: NCT06631586
Title: Standardized Microbiota Transplant Therapy in Crohn's Disease
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: GI-2024-33127
Record Dates: First submitted 2024-10-06; First posted 2024-10-08 (Actual); Last update posted 2025-02-04 (Actual); Status verified 2025-02

CONDITIONS: Crohn Disease
MeSH Terms: conditions — Crohn Disease

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CD patients randomized to MTP-101C (Experimental)
  Interventions: Biological: MTP-101C
- CD patients randomized to MTP-101S (Experimental)
  Interventions: Biological: MTP-101S

INTERVENTIONS:
Biological: MTP-101C — MTP-101C composed of double-encapsulated freeze-dried healthy donor microbiota. The fecal microbiota is frozen in the presence of a lyoprotectant (trehalose), freeze-dried, and double encapsulated into hypromellose capsules (Lonza, Morristown, NJ). Each capsule contains ≥ 1 x 10 11 and ≤ 2.0 x 10 11 bacterial cells.
  Arms: CD patients randomized to MTP-101C
Biological: MTP-101S — MTP-101S contains identical healthy donor microbiota double encapsulated in VCaps Plus (Lonza). These capsules are also composed of hypromellose but disintegrate in the proximal small bowel. Each capsule contains ≥ 1 x 10 11 and ≤ 2.0 x 10 11 bacterial cells.
  Arms: CD patients randomized to MTP-101S

SUMMARY:
Crohn's disease (CD) develops because of a disruption of homeostasis between the gut microbiota and the host immune system resulting in excessive inflammation in the intestinal tract. Current drug therapies for CD are directed at the immune system. The emergence of fecal microbiota transplantation (FMT) for the treatment of recurrent C. difficile infections (rCDI) has opened a frontier of restorative therapies targeting the gut microbiome. This study aims to assess if two forms of encapsulated FMT material (MTP101C and MTP101S) can effectively engraft in the ileum and colon of individuals with CD. This study will also assess how the impact of CD phenotype impacts engraftment. Finally this study will explore symptom and endoscopic changes before and after these two therapies.

ELIGIBILITY:
Inclusion Criteria:

* Able and willing to provide informed consent.
* 18-89 years of age.
* English speaking.
* Diagnosis of CD based on typical clinical and histologic features.
* Active disease on endoscopy:

  * SES-CD >= 6
  * SES-CD >= 4 for isolated ileal disease
* Current CD therapies are in the maintenance phase of dosing at the time of randomization.
* Any ongoing CD therapy (apart from steroid use) must be at stable doses for 4 weeks prior to randomization and remain stable over study course.
* Steroid use 20mg or less by 5 days prior to randomization.
* Steroid use stipulations:
* Prednisone must be tapered below 20mg after 7 days.
* Any use of budesonide over the study period is allowed although tapering is encouraged.
* Rescue medications: Steroid courses (up to 40mg for two weeks with a planned taper) are allowed at the discretion of the treating provider. Study drug therapy will be stopped on a case-by-case basis on discussion with the participant and treating provider.
* Women who are not post-menopausal (at least 12 months of non-therapy induced amenorrhea) or surgically sterile (e.g., absence of ovaries and/or uterus) must remain abstinent or use a highly effective form of birth control (e.g., oral contraception, transdermal patch, barrier, intrauterine device).

  o Periodic abstinence and early withdraw are not acceptable methods.
* Able to comply with study measures in the opinion of the investigator.

Exclusion Criteria:

* Extensive bowel resection: i.e., subtotal colectomy or substantial removal of small bowel where short bowel syndrome could be a concern.
* Documented gastroparesis
* History of pylorus non-preserving gastric surgery, e.g., Roux-en-Y gastric bypass.
* Symptomatic stricture defined as a stricture that:

  * Cannot be traversed by the colonoscope,
  * Requires intervention to be traversed,
  * Is otherwise responsible for the predominant clinical picture, in the opinion of the investigator.
* Presence of ileostomy or colostomy.
* Entero-vesicular fistula (i.e., fistula from bowel to bladder).
* Suspicion of ischemic colitis, radiation colitis or microscopic colitis.
* Diagnosis of ulcerative colitis.
* Active or untreated infection.
* Adenomatous polyps that have not been removed.
* Use of antibiotics within 14-days of randomization.
* Current pregnancy.
* Current breastfeeding or planning to breastfeed over the study period.
* History of anaphylactic food allergies.
* End stage liver disease or cirrhosis.
* Anticipated need for antibiotics over the study period.
* Anticipated surgical procedure over the study period.
* An absolute neutrophil count <500 cell/µL.
* Diagnosis of a primary immunodeficiency.
* Active malignancy requiring the use of chemotherapeutic agent (except for localized non-melanomatous skin cancers).
* Patients receiving active cytotoxic therapy for solid tumors and hematologic malignancies.
* Any solid organ transplant within 6 months of randomization.
* Use of chimeric antigen receptor T-cell therapy or hematopoietic cell transplant within the past 12 months
* Life expectancy >=6 months.

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2025-01-15 (Actual); Primary Completion 2029-06-15 (Estimated); Study Completion 2029-06-15 (Estimated)

PRIMARY OUTCOMES:
donor microbial engraftment | 2months
  measured in intestinal ileal biopsies

SECONDARY OUTCOMES:
Changes in ileal microbial composition | 2 months
  biopsy samples, between baseline and 2 months
Colonic engraftment of donor microbiota | 2 months
  colonic biopsies
Changes in colonic microbial composition | 2 months
Engraftment | 2 months
  measured by fecal samples over the study period.
Microbial compositional changes | 2 months
Changes in clinical symptoms | baseline, 2 months, 6 months
  measured by the Crohn's Disease Activity Index (CDAI) at baseline, 2-months, and 6-months.
Endoscopic changes in inflammation | 2 months
  measured by the Single Endoscopic Score for Crohn's Disease (SES-CD) at baseline and 2-months.
Safety and tolerability of MTT | 2 months
  measured by the rate of AEs and SAEs.

CONTACTS AND LOCATIONS:
Overall Officials: Byron Vaughn, Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States